CLINICAL TRIAL: NCT04097717
Title: Developing and Testing a Decision Support Tool for Women Making Tubal Sterilization Decisions
Brief Title: "My Decision" Tubal Sterilization Decision Support Tool
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: University of Tennessee (Other); University of California, San Francisco (Other); National Institute on Minority Health and Health Disparities (NIMHD) (NIH)
Responsible Party: Principal Investigator, Elizabeth Mosley, Professor, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: STUDY20110382; R01MD011678-01 (NIH)
Record Dates: First submitted 2019-09-19; First posted 2019-09-20 (Actual); Last update posted 2024-11-01 (Actual); Status verified 2024-10

CONDITIONS: Tubal Sterilization; Women's Health; Contraception; Contraception Behavior; Reproductive Behavior
Keywords: Tubal Ligation; Decision Aid
MeSH Terms: conditions — Contraception Behavior; Reproductive Behavior

STUDY DESIGN:
Intervention Model Description: This study is a randomized controlled trial in which participants will be assigned to one of two groups (intervention arm or usual care arm) in parallel for the duration of the study. All participants will be asked to complete assessments at three separate time points [immediately after using the decision aid (for those in the intervention arm) when participants are less than 24 weeks gestation (Time 1); in the 3rd trimester between 32-36 weeks gestation (Time 2); and three months postpartum (Time 3)].
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Decision Aid Arm (Experimental): Participants will use the web-based decision aid plus usual medical care.
  Interventions: Behavioral: "My Decision" tubal sterilization decision aid; Other: Usual Care
- Usual Care Arm (Other): Participants will receive usual medical care.
  Interventions: Other: Usual Care

INTERVENTIONS:
Behavioral: "My Decision" tubal sterilization decision aid — The "My Decision" tubal sterilization decision aid is a web-based decision aid designed to help women make informed decisions about tubal sterilization.
  Arms: Decision Aid Arm
Other: Usual Care — Usual medical care will vary among participants.

SUMMARY:
This study seeks to test a web-based decision support tool developed to enhance low-income women's ability to make informed decisions about tubal sterilization that align with their preferences, values and reproductive goals. Half of participants will receive usual care, while the other half will use the web-based decision aid plus usual care. The investigators hypothesize that compared to women who receive usual care alone, women randomized to the decision aid arm will have greater knowledge about sterilization and alternative options, lower decisional conflict, and will be more satisfied with their contraceptive decision at 3-month follow-up.

DETAILED DESCRIPTION:
Female surgical sterilization is the second most commonly used contraceptive method in the US and is disproportionately used by low-income women and women of color. Whether the higher use of sterilization in these populations reflects inappropriate overutilization is unclear. On one hand, low-income and racial minority women frequently misunderstand the permanent nature of sterilization, are often unaware of reversible contraceptive alternatives, and commonly experience regret after the procedure- suggesting suboptimal decision making. On the other hand, there is evidence of substantial unmet demand for sterilization among low-income women, due to unique access barriers posed by Medicaid sterilization regulations, putting them at high risk for unintended pregnancy and the adverse health and social consequences associated with unintended pregnancy.

Medicaid sterilization policy currently requires that all women requesting a federally-funded procedure complete a standardized consent form at least 30 days prior to sterilization. This policy was originally instituted in the 1970s to protect vulnerable women from coercive sterilization practices by attempting to ensure informed and voluntary consent. However, there is growing consensus that the policy is incapable of ensuring informed consent, and that the mandatory 30-waiting period impedes access to desired sterilization for many low-income women. The lack of a process that can ensure both informed consent and timely access for sterilization procedures hampers progress toward reproductive health equity for low-income women.

This study seeks to test a novel, web-based decision support tool to support low-income women's ability to make informed and value-concordant decisions about surgical sterilization. A decision support tool may be particularly useful in the context of sterilization decisions because this is a preference-sensitive decision with permanent implications and because there is a high level of misunderstanding about sterilization and limited awareness of alternative options among women who have undergone the surgery, indicating critical gaps in the quality of pre-sterilization counseling. Furthermore, patient-provider interactions may be complicated by a broader social and historical context in which poor and minority women's reproductive choices have not always been valued.

The study is a multi-site randomized controlled trial to test the effect of the decision aid plus usual care compared to usual care alone on decision quality among 350 racially-diverse, low-income pregnant women considering a post-partum sterilization procedure. Participant surveys will be utilized at three assessments points to evaluate outcomes.

In addition to its potential clinical utility, this research also has important policy implications, as it can inform ongoing efforts to transform the current Medicaid policy by offering a decision aid that is able to ensure informed decision making in vulnerable populations, thereby allowing the investigators to ultimately replace the current Medicaid consent form with this scalable tool. Once there is a tool to safeguard women with an evidence-based process for ensuring informed consent, further progress can be made in potentially shortening or waiving the mandatory 30-day waiting period that has restricted access to desired sterilization for many low-income women.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women
* 21-45 years of age
* Fluently speak English or Spanish
* Fluently read English or Spanish
* Considering tubal sterilization
* < 24 weeks gestation
* Continuing current pregnancy
* Using Medicaid insurance

Exclusion Criteria:

* Unable to consent to study participation
* Unable to interact with the content of the web-based decision aid

Ages: 21 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Male and Trans Male participants will not be eligible for participation in this study.
Enrollment: 549 (Actual)
Dates: Start 2020-02-24 (Actual); Primary Completion 2023-01-06 (Actual); Study Completion 2024-04-30 (Actual)

PRIMARY OUTCOMES:
Participant Knowledge about Tubal Sterilization | Less than 24 weeks gestation (Time 1)
  Participant responses to 10 True/False items adapted from previously published studies of tubal sterilization knowledge and informed by in-depth interviews with women about sterilization decision making. Items assess knowledge about tubal sterilization and alternative contraception options and will be coded as correct vs. incorrect, with "Don't Know" being coded as an incorrect response. The percentage of correct responses across the 10 questions will be calculated for each participant. The score range is 0 to 100%.
Participant Decisional Conflict in Postpartum Contraceptive Choice | Less than 24 weeks gestation (Time 1)
  Assessed by participant responses to the low literacy version of the Decisional Conflict Scale (DCS). The DCS is a validated measure to assess participants' decisional conflict in medical decision-making. The DCS low literacy version includes 10 items about experience of conflict, with "Yes" = 0, "unsure" = 2 and "No" = 4. All 10 items are a) summed; b) divided by 10; and c) multiplied by 25. Scores range from 0 (no decisional conflict) to 100 (extremely high decisional conflict).

SECONDARY OUTCOMES:
Contraceptive Method Selected | Less than 24 weeks gestation (Time 1)
  Will determine the proportion of women who select sterilization versus another method of contraception at Time 1. Assessed by participant responses to an item asking which contraceptive method they are planning to use after delivery.
Participant Satisfaction with Decision Making | Three months postpartum (Time 3)
  Assessed by participant responses to the Satisfaction with Decision Scale (SWD), a validated 6-item scale measuring participants' satisfaction with healthcare decision making. The SWD uses a 5-point Likert scale where 1 is "Strongly Disagree" and 5 is "Strongly Agree." A summary score is calculated as an average of all items with a range of 1-5, with a higher score reflecting a higher level of satisfaction with the decision.

OTHER OUTCOMES:
Participant Knowledge about Tubal Sterilization | 32-36 weeks gestation (Time 2)
  Participant responses to 10 True/False items adapted from previously published studies of tubal sterilization knowledge and informed by in-depth interviews with women about sterilization decision making. Items assess knowledge about tubal sterilization and alternative contraception options and will be coded as correct vs. incorrect, with "Don't Know" being coded as an incorrect response. The percentage of correct responses across the 10 questions will be calculated for each participant. The score range is 0 to 100%. Participant knowledge will be measured at Time 2 to assess the sustained impact of the decision aid on knowledge.
Participant Decisional Conflict in Postpartum Contraceptive Choice | 32-36 weeks gestation (Time 2)
  Assessed by participant responses to the low literacy version of the Decisional Conflict Scale (DCS). The DCS is a validated measure to assess participants' decisional conflict in medical decision-making. The DCS low literacy version includes 10 items about experience of conflict, with "Yes" = 0, "unsure" = 2 and "No" = 4. All 10 items are a) summed; b) divided by 10; and c) multiplied by 25. Scores range from 0 (no decisional conflict) to 100 (extremely high decisional conflict). Decisional conflict will be measured at Time 2 to assess the sustained impact of the decision aid on decisional conflict.
Contraceptive Method Selected | 32-36 weeks gestation (Time 2)
  Will determine the proportion of women who select sterilization versus another method of contraception at Time 2. Assessed by participant responses to an item asking which contraceptive method they are planning to use after delivery.
Contraceptive Method(s) Used | Three months postpartum (Time 3)
  Assessed by participant responses to a multiple choice item asking which methods of contraception they have used or received since their pregnancy ended.
Ease in Contraceptive Decision Making | Less than 24 weeks gestation (Time 1)
  Assessed by participant responses to a 10 point scale about ease of decision making with regards to contraceptive method selection. Response options range from 0 ("Strongly Disagree" that this is an easy decision to make) to 10 ("Strongly Agree" that this an easy decision to make").
Ease in Contraceptive Decision Making | 32-36 weeks gestation (Time 2)
  Assessed by participant responses to a 10 point scale about ease of decision making with regards to contraceptive method selection. Response options range from 0 ("Strongly Disagree" that this is an easy decision to make) to 10 ("Strongly Agree" that this an easy decision to make").
Certainty about Tubal Sterilization Decision | Less than 24 weeks gestation (Time 1)
  Assessed by participant responses to a 10 point scale indicating certainty in desire to obtain or not obtain a tubal sterilization. Response options range from 0 ("Very Certain that I Do Not Want") to 10 ("Very Certain that I Do Want").
Certainty about Tubal Sterilization Decision | 32-36 weeks gestation (Time 2)
  Assessed by participant responses to a 10 point scale indicating certainty in desire to obtain or not obtain a tubal sterilization. Response options range from 0 ("Very Certain that I Do Not Want") to 10 ("Very Certain that I Do Want").
Participant Satisfaction with Current Contraceptive Method(s) | Three months postpartum (Time 3)
  Assessed by participant responses to a 5-point Likert scale regarding satisfaction with current contraceptive method(s). Response options range from 1 ("Very Unsatisfied") to 5 ("Very Satisfied").
Participant Confidence in Contraceptive Method Selection | Three months postpartum (Time 3)
  Assessed by participant responses to a 5-point Likert scale regarding participant confidence that the method(s) is/are "right for me". Response options range from 1 ("Not at All Confident") to 5 ("Completely Confident").
Number of Pregnancies Since Delivery | Three months postpartum (Time 3)
  Assessed by participant-reported survey responses to a Yes/No item about whether a pregnancy has occurred since delivery.
Participant Satisfaction with Sterilization Counseling | Three months postpartum (Time 3)
  Participant responses to an 8-item patient-provider communication scale created by the PI to assess participant satisfaction with the sterilization counseling experience. Response options range from 1 ("Strongly Disagree") to 5 ("Strongly Agree"). Items will be examined individually. In addition, a summary score will be created with items 2,3,6 reverse coded such that the range will be 8-40 with a higher score reflecting greater satisfaction with sterilization counseling.

CONTACTS AND LOCATIONS:
Overall Officials: Sonya Borrero, MD MS, Principal Investigator — University of Pittsburgh; Elizabeth Mosley, PhD MPH, Principal Investigator — University of Pittsburgh
Locations (2):
- United States (2):
  - University of California, San Francisco, San Francisco, California
  - University of Tennessee, Knoxville, Tennessee

IPD SHARING:
Plan to Share IPD: Yes
De-identified participant data will be used for publication.
Time Frame: Publication of results will occur upon completion of the study.
Access Criteria: De-identified participant data will be used for publication.

REFERENCES:
- [Derived] Borrero S, Mosley EA, Wu M, Dehlendorf C, Wright C, Abebe KZ, Zite N. A Decision Aid to Support Tubal Sterilization Decision-Making Among Pregnant Women: The MyDecision/MiDecision Randomized Clinical Trial. JAMA Netw Open. 2024 Mar 4;7(3):e242215. doi: 10.1001/jamanetworkopen.2024.2215. PMID 38502127